CLINICAL TRIAL: NCT05878964
Title: Evaluation of Skin Health and Quality of Life in Patients Receiving Anticancer Therapies Based on Monoclonal Antibody Anti-PD1/PDL1/CTLA4 or Cyclin-dependent Kinase (CDK) Inhibitors
Brief Title: Evaluation of Skin Health and QoL in Pts Receiving Anti-PD1/PDL1/CTLA4 or CDK Inhibitors.
Acronym: SkinHealth
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5455
Record Dates: First submitted 2023-05-08; First posted 2023-05-30 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer; Breast Cancer; Kidney Cancer; Bladder Cancer; Gastric Cancer; Skin Cancer; Melanoma; Head Neck Cancer
Keywords: immunotherapy; cyclin-dependent kinase (CDK) inhibitors; cutaneous toxicity
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Kidney Neoplasms; Urinary Bladder Neoplasms; Stomach Neoplasms; Skin Neoplasms; Melanoma; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: All patients affected by solid tumors already in treatment with anti-PD1/PDL1 or cyclin-dependent kinase (CDK) inhibitors.
  Interventions: Other: EQ-5D-5L questionnaire; Other: FACT-G (Functional Assessment of Cancer Therapy - General); Other: FACT-EGFRI-18 (Functional Assessment of Cancer Therapy - Epidermal Growth Factor Inhibitors 18 Item)
- Group 2: All patients affected by solid tumors already eligible for treatment with anti-PD1/PDL1 or cyclin-dependent kinase (CDK) inhibitors.
  Interventions: Other: EQ-5D-5L questionnaire; Other: FACT-G (Functional Assessment of Cancer Therapy - General); Other: FACT-EGFRI-18 (Functional Assessment of Cancer Therapy - Epidermal Growth Factor Inhibitors 18 Item)

INTERVENTIONS:
Other: EQ-5D-5L questionnaire — Quality of life evaluation questionnaire
Other: FACT-G (Functional Assessment of Cancer Therapy - General) — Quality of life evaluation questionnaire
Other: FACT-EGFRI-18 (Functional Assessment of Cancer Therapy - Epidermal Growth Factor Inhibitors 18 Item) — Self reported evaluation of cutaneous toxicity questionnaire.

SUMMARY:
The study aim to investigate the relationship between cutaneous adverse events and quality of life in patients taking immune check point inhibitor or cyclin-dependent kinase (CDK) 4 and 6 inhibitors by two steps. In the first one, it will be investigated the relationship between the skin toxicity related to the use selected therapies and the quality of life of patients already receiving these therapies for treatment of their cancer. In the second one, it will be evaluated the relationship between skin toxicity and quality of life over three months of treatment in patients initially naïve for selected therapies. Cancer included in the analysis are NSCLC, renal cancer, gastric cancer, breast cancer, bladder cancer, melanoma, squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

(for all Groups)

1. Age ≥ 18 years.
2. Histological diagnosis of solid tumor.
3. Patient able to complete the questionnaires submitted during the study.
4. Signed written informed consent. (for Group I) Patients already under treatment for at least three months with anti-PD1/PDL1/ CTLA4 or cyclin-dependent kinase (CDK) inhibitors for any type of cancer. Treatment considered for each cancer are only those approved by AIFA for each tumor.

(for Group II) Patients eligible for treatment with anti-PD1/PDL1/ CTLA4 or cyclin-dependent kinase (CDK) inhibitors for any type of cancer. Treatment considered for each cancer are only those approved by AIFA for each tumor.

Exclusion Criteria (for all Groups):

1. Age < 18 y.o.
2. Skin diseases or alterations present before the beginning of anti-PD1/PDL1 or cyclin-dependent kinase (CDK) inhibitors.
3. Chronic use of steroids.
4. Previous psychiatric disorders or patients taking antidepressant.
5. Refusal to sign written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients affected by solid tumors already in treatment (Phase I) or eligible for treatment (Phase II) with anti-PD1/PDL1 or cyclin-dependent kinase (CDK) inhibitors at the unit of Medical Oncology of Fondazione Policlinico Universitario Agostino Gemelli IRCCS of Rome for any type of cancer, and satisfying the related inclusion criteria onwards exposed.
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Quality of life in patients undergoing anti-PD1/PDL1/CTLA4 or cyclin-dependent kinase (CDK) inhibitors evaluated by EQ-5D-5L questionnaire. | 18 months
  To evaluate the correlation between skin toxicity and quality of life over three months of treatment in patients initially naïve for monoclonal antibody anti-PD1/PDL1/CTLA4 or with cyclin-dependent kinase (CDK) inhibitors.
  Skin toxicity will be evaluated by the physician and graded based ob CTCAE v 5.0.
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Quality of life during therapy with anti-PD1/PDL1/CTLA4 or cyclin-dependent kinase (CDK) inhibitors by FACT-G scale | 18 months
  To evaluate the correlation between skin toxicity and quality of life over three months of treatment in patients initially naïve for monoclonal antibody anti-PD1/PDL1/CTLA4 or with cyclin-dependent kinase (CDK) inhibitors.
  Skin toxicity will be evaluated by the physician and graded based ob CTCAE v 5.0.
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. For all FACIT measures, higher scores are better than lower scores.
Quality of life during therapy with anti-PD1/PDL1/CTLA4 or cyclin-dependent kinase (CDK) inhibitors by FACT-EGFRI-18 scale. For all FACIT measures, higher scores are better than lower scores. | 18 months
  To evaluate the correlation between skin toxicity and quality of life over three months of treatment in patients initially naïve for monoclonal antibody anti-PD1/PDL1/CTLA4 or with cyclin-dependent kinase (CDK) inhibitors.
  Skin toxicity will be evaluated by the physician and graded based ob CTCAE v 5.0.

SECONDARY OUTCOMES:
Role of gender | 18 months
  To describe differences in quality of life based on gender. The incidence and grade of skin toxicity based ob CTCAE v 5.0, will be estimated based on sex. Similarly the correlation of skin toxicity with quality of life evaluated by EQ-5D-5L, FACT-G, FACT-EGFRI-18 measures will be estimated by sex.
Role of therapy | 18 months
  To describe differences in quality of life based on type of therapy received (Immunotherapy vs CDK inhibitors).
  The incidence and grade of skin toxicity based ob CTCAE v 5.0, will be estimated based on type of therapy. Similarly the correlation of skin toxicity with quality of life evaluated by EQ-5D-5L, FACT-G, FACT-EGFRI-18 measures will be estimated by type of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Iacovelli, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Roberto Iacovelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No